CLINICAL TRIAL: NCT04009980
Title: Long-term Morphological and Functional Retinal Changes After Topical Citicoline Administration in Patients With Mild Signs of Diabetic Retinopathy in Type 1 Diabetes Mellitus: Pilot Study
Brief Title: Long-term Retinal Changes After Topical Citicoline Administration in Patients With Mild Signs of Diabetic Retinopathy in Type 1 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Mariacristina Parravano, Head of Retina Unit, Fondazione G.B. Bietti, IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RET04/2015
Record Dates: First submitted 2019-06-06; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Retinopathy
Keywords: citicoline; neuropathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, randomized, double-masked, monocentric pilot study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMK2 group (Experimental): Patients receiving topical administration of OMk2 ophthalmic solution for 36 months three times/day
  Interventions: Other: OMK2 group
- Placebo group (Placebo Comparator): Patients receiving receiving only the excipients of OMk2 (placebo) for 36 months three times/day
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: OMK2 group — topical administration of OMk2 ophthalmic solution for 36 months three times/day
  Arms: OMK2 group
Other: Placebo group — topical administration of ophthalmic placebo solution for 36 months three times/day
  Arms: Placebo group

SUMMARY:
Citicoline (cytidine-5'-diphosphocholine) is an essential precursor in the synthesis of phosphatidylcholine, a component of cell membranes. Several experimental in vitro and in vivo studies have suggested that citicoline plays a neuroprotective role.

A recent clinical study has shown that treatment with topical citicoline induces, after 60 days of therapy, a significant improvement in the ganglion cell function .In addition topical citicoline has been demonstrated in vivo a neuroprotective effect in preventing diabetic retinopathy .

The Investigators want to evaluate if citicoline may reduce the progression of retinal damage in patients with mild diabetic retinopathy.

DETAILED DESCRIPTION:
The investigators evaluated patients with mild signs of diabetic retinopathy (DR) treated with eye-drop solution with citicoline ( OMk2 ophthalmic solution).

All patients was randomized in two groups (10:10), one receiving topical administration of OMk2 ophthalmic solution for 36 months and one group receiving only the excipients of OMk2 (placebo).

Omk2 ophthalmic solution and the placebo will be used for 36 months three times/day.

They will undergo a complete ocular examination at baseline and at 6-, 12-, 18-, 24-, 30- and 36- months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 DM
* Diagnosis of mild Diabetic rethnopathy (DR)
* Retinal sensitivity impairment evaluated by means of frequency doubling technology (Matrix FDT) with a mean deviation (MD) p value <5% or with two locations with p <5% and one location with p<1% in the total or pattern deviation plots.

Exclusion Criteria:

* Hyperopia higher than +5 diopter (D)
* myopia higher than -8 D
* astigmatism higher than 2 D
* Visual acuity below 20/25
* significant media opacity
* previous ocular surgery
* previous diagnosis of glaucoma
* uveitis
* retinal disease other than mild diabetic retinopathy
* patients with any ocular disease
* systemic disease other than diabetes
* Any signs of diabetic retinopathy more advanced than mild as coded by ICDRSS (e.g. macular edema or any sign of proliferative DR)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Changes of Retinal sensitivity and contrast sensitivity function after topical citicoline use in patients with diabetic retinopathy | Functional retinal changes at 36 months
  To evaluate functional retinal parameters : retinal sensitivity by Humphrey Matrix and contrast sensitivity function by Pelli Robson in patients with diabetic retinopathy

SECONDARY OUTCOMES:
Morphological retinal changes after topical citicoline use in patients with diabetic retinopathy | Morphological retinal changes at 36 months
  To evaluate morphological retinal parameters by Spectral Domain OCT( SD-OCT ) and by Adaptive Optics (AO) at each time point of follow up : retinal thickness, RNFL thickness, inner retinal thickness and outer retinal thickness.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione G.B.Bietti, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Dijk HW, Verbraak FD, Kok PH, Garvin MK, Sonka M, Lee K, Devries JH, Michels RP, van Velthoven ME, Schlingemann RO, Abramoff MD. Decreased retinal ganglion cell layer thickness in patients with type 1 diabetes. Invest Ophthalmol Vis Sci. 2010 Jul;51(7):3660-5. doi: 10.1167/iovs.09-5041. Epub 2010 Feb 3. PMID 20130282
- [Background] Vujosevic S, Midena E. Retinal layers changes in human preclinical and early clinical diabetic retinopathy support early retinal neuronal and Muller cells alterations. J Diabetes Res. 2013;2013:905058. doi: 10.1155/2013/905058. Epub 2013 Jun 12. PMID 23841106
- [Background] Diederich K, Frauenknecht K, Minnerup J, Schneider BK, Schmidt A, Altach E, Eggert V, Sommer CJ, Schabitz WR. Citicoline enhances neuroregenerative processes after experimental stroke in rats. Stroke. 2012 Jul;43(7):1931-40. doi: 10.1161/STROKEAHA.112.654806. Epub 2012 May 10. PMID 22581817
- [Background] Parisi V, Coppola G, Centofanti M, Oddone F, Angrisani AM, Ziccardi L, Ricci B, Quaranta L, Manni G. Evidence of the neuroprotective role of citicoline in glaucoma patients. Prog Brain Res. 2008;173:541-54. doi: 10.1016/S0079-6123(08)01137-0. PMID 18929133
- [Background] Parisi V, Manni G, Colacino G, Bucci MG. Cytidine-5'-diphosphocholine (citicoline) improves retinal and cortical responses in patients with glaucoma. Ophthalmology. 1999 Jun;106(6):1126-34. doi: 10.1016/S0161-6420(99)90269-5. PMID 10366081
- [Background] Roberti G, Tanga L, Parisi V, Sampalmieri M, Centofanti M, Manni G. A preliminary study of the neuroprotective role of citicoline eye drops in glaucomatous optic neuropathy. Indian J Ophthalmol. 2014 May;62(5):549-53. doi: 10.4103/0301-4738.133484. PMID 24881599
- [Derived] Parravano M, Scarinci F, Parisi V, Giorno P, Giannini D, Oddone F, Varano M. Citicoline and Vitamin B12 Eye Drops in Type 1 Diabetes: Results of a 3-year Pilot Study Evaluating Morpho-Functional Retinal Changes. Adv Ther. 2020 Apr;37(4):1646-1663. doi: 10.1007/s12325-020-01284-3. Epub 2020 Mar 16. PMID 32180131